CLINICAL TRIAL: NCT03583255
Title: A Combination Therapy for Cancer-Related Fatigue in Advanced Cancer Patients
Brief Title: Physical Activity With or Without Dexamethasone in Reducing Cancer-Related Fatigue in Patients With Locally Advanced, Metastatic, or Recurrent Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2018-0226; NCI-2018-01103 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0226 (Other: M D Anderson Cancer Center); R21NR016737 (NIH)
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid System Neoplasm; Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (dexamethasone, exercise) (Experimental): Patients receive dexamethasone PO BID for 7 days. Patients also complete resistance training and moderate intensity walking at home for minimum 5 days per week over 4 weeks.
  Interventions: Drug: Dexamethasone; Behavioral: Exercise Intervention
- Arm II (placebo, exercise) (Active Comparator): Patients receive placebo PO BID for 7 days. Patients also complete resistance training and moderate intensity walking as in Arm I.
  Interventions: Behavioral: Exercise Intervention; Other: Placebo Administration

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm I (dexamethasone, exercise)
Behavioral: Exercise Intervention — Complete resistance training and moderate intensity walking
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo, exercise)

SUMMARY:
This phase II/III trial studies how well physical activity with or without dexamethasone works in reducing cancer-related fatigue in patients with cancer that has spread to other places in the body or has come back. Dexamethasone may decrease the body's immune response. Combining physical activity with dexamethasone may help to treat fatigue in patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypotheses that patients with cancer-related fatigue (CRF) will be satisfied with the physical activity + dexamethasone (PA+ DEX) intervention, have adequate rates of adherence, and that PA+ DEX will be feasible for patients with CRF.

Ia. To determine if the combination of PA+ DEX is a feasible intervention for advanced cancer patients, as evidenced by an adherence rate to daily use of PA+ DEX greater than or equal to 75%.

Ib. To determine if patients are satisfied with PA+ DEX, based on more than 75% of patients indicating their satisfaction with PA+ DEX with a rating of "somewhat satisfied" or "completely satisfied."

SECONDARY OBJECTIVES:

I. To test the hypothesis that PA+ DEX (PA for 4 weeks plus dexamethasone 4 mg twice a day for 1 week) will be more efficacious than PA+ placebo (PA for 4 weeks plus placebo for 1 week) on CRF as measured by the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F).

Ia. To determine if PA+ DEX results in robust reduction in FACIT-F subscale scores (defined as >= 10 point improvement in 60% of patients).

II. To explore the effects of PA+ DEX on fatigue-related symptoms and function. IIa. To determine if PA+ DEX improves CRF by targeting the various associated factors of CRF.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive dexamethasone orally (PO) twice daily (BID) for 7 days. Patients also complete resistance training and moderate intensity walking at home for minimum 5 days per week over 4 weeks.

ARM II: Patients receive placebo PO BID for 7 days. Patients also complete resistance training and moderate intensity walking as in Arm I.

After completion of study, patients are followed up at 29 days and 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced cancer (defined as metastatic or recurrent cancer or completed 2 lines of therapy) with fatigue >= 4/10 (0-10 scale) on the Edmonton Symptom Assessment Scale (ESAS)
* Presence of fatigue for at least 2 weeks
* Normal cognition defined as Memorial Delirium Assessment Scale (MDAS) of =< 13/30 completed in person or via video conference
* Hemoglobin > 8 g/L within 2 weeks of enrollment in the study
* Zubrod performance status =< 2
* Life expectancy of >= 4 months
* Able to read, write, and speak English

Exclusion Criteria:

* Patients with a history of hypersensitivity to dexamethasone or having any contraindication to physical activity as determined by the treating physician
* Reports of a fall in the past 30 days
* Uncontrolled diabetes mellitus as defined by a random blood sugar of > 200 mg/dl not being monitored by their primary care physician
* Sepsis and/or acute, chronic, or ongoing infections that are currently being treated with systemic antimicrobials
* Current, active peptic ulcer disease
* Neutropenia as defined by an absolute neutrophil count (ANC) of < 1000 cells/mm
* Regular participation in moderate- or vigorous-intensity physical activity for >= 30 minutes at least 5 times a week and strength training for >= 2 days
* Symptomatic cardiac disease (New York Heart Association functional class III or IV) or coronary artery disease
* Patients currently on immunotherapy
* Inability to comply with study protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility For Participants with Cancer-Related Fatigue (CRF) | Up to 1 month
  Will be assessed by the proportion of participants completing the intervention. Will estimate 95% confidence intervals for the proportion of patients completing the intervention.
Adherence | Up to 1 month
  Will be calculated as the mean of the % of total prescribed strength training sessions and the % of total prescribed walking regimen minutes completed (exercise), and mean (across all patients) percentage of total prescribed pills taken (study medication) as detailed above. Will estimate 95% confidence intervals for the proportion of patients completing the intervention and the adherence rate.
Satisfaction | Up to 1 month
  Will estimate 95% confidence intervals for the proportion of patients with a satisfaction rating of "somewhat satisfied" or "completely satisfied."

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yennurajalingam S, Valero V, Smalgo BG, Overman MJ, Dasari A, Wolff RA, Raghav KPS, Barcenas CH, Busaidy NL, Fellman B, Basen-Engquist K, Hess KR, Tripathy D, Bruera E. Physical Activity and Dexamethasone for Cancer-Related Fatigue: A Preliminary Placebo-Controlled, Randomized, Double-Blind Trial. J Natl Compr Canc Netw. 2025 Jan 7;23(1):e247071. doi: 10.6004/jnccn.2024.7071. PMID 39773433
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org